CLINICAL TRIAL: NCT06427044
Title: Effect of Bupivacaine Liposome Anterior Serratus Deep Block on Chronic Pain After Breast Cancer Surgery: a Randomized Controlled Study
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Lu Hua (Other)
Responsible Party: Sponsor-Investigator, Lu Hua, Assistant Professor, Tongji Hospital
Organization: Tongji Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TJ-IRB202403018
Record Dates: First submitted 2024-05-19; First posted 2024-05-23 (Actual); Last update posted 2024-05-23 (Actual); Status verified 2024-05

CONDITIONS: Breast Cancer Patients With Chronic Pain After Surgery

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Anterior serratus block group (Experimental): Bupivacaine lipid 20mL (20mL 266mg bupivacaine liposomes) was ultrasound-guided for a single anterior serranus plane block
  Interventions: Drug: Anterior serratus block group
- Control group (No Intervention)

INTERVENTIONS:
Drug: Anterior serratus block group — Bupivacaine lipid 20mL (20mL 266mg bupivacaine liposomes) was ultrasound-guided for a single anterior serranus plane block
  Arms: Anterior serratus block group

SUMMARY:
This study aims to investigate the effect and influence of liposome bupivacaine anterior serrat plane block on postoperative chronic pain in breast cancer patients, evaluate the therapeutic effect of liposome bupivacaine in postoperative chronic pain, and provide a new method for patients with postoperative chronic pain.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (aged ≥18 years) who are scheduled to undergo unilateral modified radical breast cancer surgery

Exclusion Criteria:

* 1. Patients with coagulation dysfunction 2. There are infected patients at the puncture site 3. For patients allergic to any trial drug 4. Patients who take painkillers within 48 hours before surgery 5. Severe cardiopulmonary insufficiency, such as EF< 40%, FEVC < 50% expected; Uncontrolled hypertension; 6. Refuse to perform nerve block puncture 7. Mental disorders, epilepsy history; 8. Unable to give informed consent or are participating in other clinical trials.

Ages: 18 Years to 70 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 143 (Estimated)
Dates: Start 2024-05-25 (Estimated); Primary Completion 2024-12-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of chronic pain 3 months after surgery | Three months after surgery
  Pain levels were measured three months after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Tongji Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No